CLINICAL TRIAL: NCT04479384
Title: The Immediate Effect of an Osteopathic Manual Treatment on Blood Pressure in Adults With Hypertension - a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Academy of Osteopathy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201910 EN PEDERSEN M PROTOCOL
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: High Blood Pressure
Keywords: Hypertension; Manual techniques; Blood Pressure; Osteopathy; Treatment
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Thoracic manipulation T1-T5 if somatic dysfunction. Intrathoracic fascia stretch x 3. Recoil sternum x 3. Cranial base release - 4 steps.
  Interventions: Other: Manual therapy - osteopathic techniques
- Control group (No Intervention): Supine position 10 minutes on the bench.

INTERVENTIONS:
Other: Manual therapy - osteopathic techniques — * HVLAT if any somatic dysfunction in T1-T5
  * Stretch intrathoracic fascia x 3
  * Recoil sternum x 3
  * Cranial base release, 4 phases
  Arms: Intervention group

SUMMARY:
The aim of this study was to determine if 4 manual osteopathic treatment techniques; Spinal manipulation, stretch intrathoracic fascia, sternum recoil and cranial base release has an immediate effect on blood pressure (BP) in hypertensive adults.

DETAILED DESCRIPTION:
30 hypertensive adults (age=50.76±8.66 years, height= 1.75±0.082 m, weight=89.5±19.08 kg), were randomly assigned into one of two equally sized groups; a non- intervention and an intervention group in which patients received 4 manual techniques. Outcome measures included systolic- and diastolic BP pre-treatment and post-treatment 1-,5-, and 10-minutes. Two-way mixed ANOVA was used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-60 years old.
* Primary hypertension.
* Hypertension not more than grade 2, defined as: Systolic BP from 135-174 mmHg and diastolic BP from 85-104 mmHg.

Exclusion Criteria:

* Hypertension grade 3, defined as: Systolic BP from >175 mmHg and diastolic BP >105 mmHg, due to high risk of developing stroke, apoplexy and myocardial infarct.
* Positive hepato-jugular-reflux test, as a safety-test, to test pathological conditions of the heart.
* History of liver, kidney or known heart diseases, diagnosed by family physician as these conditions can contribute to secondary hypertension.
* Presence of contraindications for manual treatment, such as (but not limited to); infections, neurological symptoms, inflammation, haemophilia, ankylosis, prosthesis, pregnancy, cancer, osteoporosis, trauma and the use of blood-thinning medicines or corticosteroids.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure baseline | Baseline
  Systolic blood pressure and diastolic blood pressure
Systolic and diastolic blood pressure post 1-minute | Post 1-minute
  Systolic blood pressure and diastolic blood pressure
Systolic and diastolic blood pressure post 5-minute | Post 5-minute
  Systolic blood pressure and diastolic blood pressure
Systolic and diastolic blood pressure post 10-minute | Post 10-minute
  Systolic blood pressure and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Mette Pedersen, BSc, Principal Investigator — International Academy of Osteopathy
Locations (1):
- Næstved Rygcenter, Næstved, Denmark